CLINICAL TRIAL: NCT03885713
Title: Identification of Predictive Biomarkers for Response to Biologic Therapies and Tofacitinib in Inflammatory Bowel Disease by Proteomic and Mass Cytometry Approaches
Brief Title: Identification of Predictive Biomarkers for Response to Biologic Therapies and Tofacitinib in Inflammatory Bowel Disease
Acronym: BioIBD
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Fundación de Investigación Biomédica - Hospital Universitario de La Princesa (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GIS-2018-BioIBD
Record Dates: First submitted 2019-03-04; First posted 2019-03-22 (Actual); Last update posted 2025-03-17 (Actual); Status verified 2025-03

CONDITIONS: Inflammatory Bowel Diseases; Crohn Disease; Ulcerative Colitis
Keywords: inflammatory bowel diseases; Crohn Disease; Ulcerative Colitis; Infliximab; Adalimumab; Golimumab; Vedolizumab; Ustekinumab; Anti-TNF; Tofacitinib
MeSH Terms: conditions — Inflammatory Bowel Diseases; Crohn Disease; Colitis, Ulcerative | interventions — Infliximab; Adalimumab; golimumab; vedolizumab; Ustekinumab; tofacitinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Patients with treatment (Active Comparator): Infliximab (Infusion 5mg/kg milligram(s)/Kilogram-Intravenous use) per clinical practice, or adalimumab (Subcutaneus 40 mg milligram(s)) per clinical practice, or golimumab (subcutaneus 50 mg milligram(s)) per clinical practice, or vedolizumab (infusion 300 mg milligram(s)) per clinical practice or ustekinumab (subcutaneous 90 mg milligram(s)) per clinical practice or tofacitinib (oral 5mg bid oral) per clinical practice
  Interventions: Biological: Infliximab or adalimumab or golimumab or vedolizumab or ustekinumab or tofacitinib
- healthy control (No Intervention): Patients without treatment

INTERVENTIONS:
Biological: Infliximab or adalimumab or golimumab or vedolizumab or ustekinumab or tofacitinib — Infliximab (Infusion 5mg/kg milligram(s)/Kilogram-Intravenous use) per clinical practice or adalimumab (Subcutaneus 40 mg milligram(s)) per clinical practice or golimumab (subcutaneus 50 mg milligram(s)-subcutaneus) per clinical practice or vedolizumab (infusion 300 mg milligram(s)) per clinical practice or ustekinumab (subcutaneous 90 mg milligram(s)) per clinical practice or tofacitinib (oral 5mg bid)
  Arms: Patients with treatment

SUMMARY:
Prospective, multicentre trial which the biologic treatment will be initiated by clinical indication. The treatment selection anti-TNFα (infliximab, adalimumab or golimumab), vedolizumab, ustekinumab and tofacitinib will be made at the discretion of the clinician. There will be no random assignment of treatment. The drugs will be used in the approved indications and conditions of use.

DETAILED DESCRIPTION:
Background

IBD, including CD and UC, is a chronic disorder of unknown etiology that involves a pathological response of the immune system, resulting in chronic inflammation of the gastrointestinal tract. IBD generally affects young patients, being a highly disabling disease. Unfortunately IBD has no current treatment, so the therapeutic goal is to keep the inflammatory process under control in order to prevent the onset of symptoms and the development of further complications.

The complexity and costs associated with the treatment of IBD make it a very relevant disease. Specifically in the USA, where it is one of the five diseases with the greatest social burden, with an annual cost of 1,700 million dollars for health services. In Europe, the annual costs (direct and indirect) associated with IBD exceed 25,000 million euros. Together, this highlights the strategic importance of IBD for society, including both patients and the health system.

IBD prevalence is high, affecting more than 1.6 million inhabitants in the US and more than 2.2 million in Europe. On the other hand, its incidence varies widely depending on the different countries. Nevertheless, in a generalized manner, it is increasing rapidly, probably due to the "westernization" of lifestyles. Indeed, a large multicenter study leaded by the host institution suggests that the current incidence is greater than previously described.

In addition, the cost associated with IBD diagnosis and treatment is increasing over time, either because of the costs associated with the treatment itself or due to the greater complexity of the diagnostic tests and tools to which these patients are subjected.

Despite the increasingly frequent use of immunosuppressant drugs, the need for surgery due to IBD has not changed substantially in recent decades. It has been suggested that early initiation of treatment with immunosuppressants and biologics to induce remission would prevent the onset of complications of the disease. However, this widely applied strategy would lead to overtreatment of patients who would have had a benign course of the disease. On the other hand, the current treatment strategy is similar in almost all patients with IBD: it starts, in general, with the less aggressive drugs, progressively moving to more potent therapies when previous treatments have failed. In this way, the window of opportunity to prevent complications in more complex patients is often lost. Thus, because there are no prognostic factors that have proven useful in clinical practice, the selection of a treatment for each patient remains empirical, adapted according to clinical evolution and difficulties of each case.

Anti-TNFα drugs have been shown to be effective for induction of remission and maintenance thereof in patients with IBD. In 2014, the use of vedolizumab was approved, both for CD and UC, whose therapeutic targets are α4β7 integrins. In 2016, ustekinumab, directed against the p40 subunit shared by interleukins 12 and 23, was approved in patients with CD, thus increasing the therapeutic arsenal against IBD. All these biologic drugs have a high cost, so they pose a great economic burden for health systems. However, approximately only one third of patients will achieve remission. At present, the medical community does not have reliable criteria for selecting which patients will benefit from any of the above-mentioned drugs. Thus, the variables (epidemiological, clinical, analytical, etc.) usually used to predict patients' response to biological therapy have shown little utility. Therefore, it is a priority in the study of IBD the identification of those molecular and cellular pathways involved in the onset of IBD in each patient, in order to make a more rational use of resources. Achieving that goal will allow us to indicate the most appropriate treatment to each individual, hence avoiding administering drugs to patients who will not respond (which implies an inadequate use of resources and an unjustified risk of adverse effects).

The identification of biomarkers with capacity to predict clinical response to biologic drugs is, therefore, an area of great interest. In this context, "omic" techniques allow massive searches at various levels, including DNA (genomics) and its modifications (epigenome), RNA (transcriptome), proteins (proteome), bacterial composition (microbiome), etc. This project aims to deepen this aspect through the use of 2 massive last-generation approaches that will identify the signaling routes (proteomics) and the immune cell subsets (mass cytometry) involved in the response to biologic drugs. This will ultimately lead to the identification, in an unbiased manner, of novel predictive biomarkers for response to biologic therapies in IBD.

Study population

* Group 1: Patients with IBD that will start treatment with a biologic drug or tofacitinib according to medical criteria in the context of the usual clinical practice.
* Group 2: Individuals without IBD in whom an ileocolonoscopy is performed and is normal.

Definitions

Endoscopic activity:

* In patients with CD, it will be evaluated using the Simplified Endoscopic Activity Score for Crohn's Disease (SES-CD); Endoscopic activity will be considered when the SES-CD is ≥3. In operated patients, or in those where the endoscopic exploration is incomplete, the SES-CD will be calculated according to the explorable segments, considering the previously described activity criterion.
* In patients with UC, it will be evaluated by the Mayo endoscopic sub-score; endoscopic activity will be considered as ≥2.
* The assessment of endoscopic activity will be carried out centrally by sending anonymized endoscopic images.

Endoscopic response (main endpoint):

* In patients with CD, the endoscopic response will be defined as a >50% decrease in the SES-CD14 weeks after starting the biologic treatment. As a secondary variable, endoscopic response will be also defined as a decrease ≥3 points in the SES-CD (considered as a clinically significant endoscopic improvement). There is consensus that the evaluation of the response to treatment (and therefore the consideration of a patient as a primary non-responder) should not be performed before week 12-14 (in patients treated with anti-TNFα drugs).
* In patients with UC, the endoscopic response will be defined as a decrease of ≥1 point in the Mayo endoscopic sub-score 14 weeks after starting the biologic treatment.

Endoscopic remission:

* In patients with CD, endoscopic remission will be defined as a SES-CD ≤2, 14 weeks after starting the biologic treatment.
* In patients with UC, endoscopic remission will be defined as an endoscopic subscript ≤1, 14 weeks after starting the biologic treatment.

Clinical activity:

* In patients with CD, it will be evaluated using the Crohn's Disease Activity Index (CDAI). Clinical remission will be considered as a CDAI <150 points 14 weeks after starting the biologic treatment; and clinical response, reduction of CDAI by 100 (R-100) or 70 points (R-70).
* In patients with UC it will be evaluated by the partial Mayo index. Clinical remission will be considered as a partial Mayo index ≤2, with all the scores (of the partial index) of 1 as a maximum and with a sub-score of rectal bleeding of 0, 14 weeks after starting the biologic treatment; and clinical response, the decrease of 3 or more points (of the partial index) with respect to the baseline situation.

Sample size

The sample size for the laboratory analyses will be 30 in each of the subgroups of patients: 1) CD treated with anti-TNFα drugs; 2) CD treated with vedolizumab; 3) CD treated with ustekinumab; 4) UC treated with anti-TNFα; 5) UC treated with vedolizumab; 6) UC treated with tofacitinib. Since the total number of patients is 180, the inclusion for each of the 17 participating centers will be approximately 9 patients, a perfectly viable figure in the allocated timeframe. It is estimated that the percentage of endoscopic response (primary endpoint) is 30% so in each subgroup there will be 10 responding patients and 20 patients with treatment failure, an adequate number for the evaluation of biomarkers predictors of response. In addition, 30 healthy controls will be included to compare the obtained results in the IBD patients.

Development of the study

The present study is organized in 3 visits: visit 1, prior to initiating the treatment; visit 2, at 14 weeks after starting treatment; and visit end of study. The investigators will use their proved expertise in previous clinical trials to coordinate and monitor all the research centers using the online AEG-RedCap platform. Data collection forms will be provided to all the centers prior to start the study. The overall duration of the study is estimated at 3 years (20 months of inclusion + 4 months of follow-up + 12 months for analysis).

ELIGIBILITY:
Group 1: Patients with IBD

Inclusion Criteria:

* Over 18 years.
* Diagnosis of IBD according to the criteria of the European Crohns and Colitis Organization (ECCO).
* Have indication of treatment with a biologic drug or tofacitinib.
* Be the first received drug with a given mechanism of action (anti-TNFα, anti-α4β7, anti-p40 or Janus kinase (JAK) inhibitor).
* Have endoscopic activity of IBD within 1 month of starting the biologic treatment (see definitions section: SES-CD ≥ 3 in CD and endoscopic sub-index of May ≥ 2 in UC).
* In the case of CD, receive the biologic treatment by luminal activity (not perianal).

Exclusion Criteria:

* Under 18 years old.
* Having an immune-mediated disease other than IBD at the baseline visit.
* Having a neoplasm or an active infection at the time of the baseline visit.
* Pregnancy or lactation.
* Alcohol or drug abuse.
* Ostomy.
* Abdominal surgery in the last 6 months.
* Colectomy in patients with UC.
* Active infection with hepatitis B, C or HIV virus.
* Indication of biologic treatment for a cause other than IBD.
* Indication of biologic treatment to prevent postoperative recurrence in CD.
* Have previously received a drug with the same mechanism of action of the drug indicated by your doctor (anti-TNFα, anti-α4β7, anti-p40 or JAK inhibitor).
* Refusal to give consent for participation in the study.

Group 2: patients without IBD

Inclusion Criteria:

- Patients not diagnosed with IBD, or other inflammatory, allergic, malignant or autoimmune diseases, where a ileocolonoscopy is performed due to the normal clinical practice.

Exclusion Criteria:

* Under 18 years old.
* Advanced chronic disease or any other pathology that prevents the follow-up of the protocol of this study.
* Pregnancy or lactation.
* Active infection with hepatitis B, C or HIV virus.
* Alcohol or drug abuse.
* Finding of macroscopic alterations during the ileocolonoscopy, or finding of relevant inflammatory alterations in the biopsies obtained during the ileocolonoscopy.
* Refusal to give consent for participation in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 180 (Actual)
Dates: Start 2019-09-10 (Actual); Primary Completion 2024-12-31 (Actual); Study Completion 2024-12-31 (Actual)

PRIMARY OUTCOMES:
Identify predictive tissue and blood biomarkers for response to biologic therapies and tofacitinib in Crohn´s disease and ulcerative colitis | 14 weeks
  will be calculated for each of the selected biomarkers: sensitivity, specificity, positive predictive value, negative predictive value, positive likelihood ratio and negative likelihood ratio

SECONDARY OUTCOMES:
Identify non-invasive blood biomarkers of endoscopical inflammation | 14 weeks
  will be calculated for each of the selected biomarkers: sensitivity, specificity, positive predictive value, negative predictive value, positive likelihood ratio and negative likelihood ratio
Evaluate the effect of the treatment on the immune subsets and study the signaling pathways specifically modulated | 14 weeks
  To achieve this outcome will be used endoscopic response defined in CD patients as a decrease of 50% in SES-CD(78) 14 weeks after starting treatment and defined in UC patients as a decrease ≥1 point in the mayo score (82) 14 weeks after starting treatment
Generate a collection of biological simple (Blood sample, urine sample, stool sample, biopsy simple) | 14 weeks
  these samples will be use to reach the outcomes of this study and will be used in future studies

CONTACTS AND LOCATIONS:
Overall Officials: Javier P Gisbert, Principal Investigator — Fundación de Investigación Biomédica - Hospital Universitario de La Princesa
Locations (21):
- Spain (21):
  - Hospital General Universitario de Alicante, Alicante, Alicante
  - Hospital Universitario Parc Taulí, Sabadell, Barcelona
  - Hospital Universitario Marqués de Valdecilla, Santander, Cantabria
  - Hospital Público General de Tomelloso, Tomelloso, Ciudad Real
  - Hospital Universitario Reina Sofía, Córdoba, Córdoba
  - Hospital Universitario Donostia, Donostia / San Sebastian, Donostia
  - Hospital Universitario Dr. Josep Trueta, Girona, Gerona
  - Hospital Juan Ramón Jiménez, Huelva, Huelva
  - Hospital San Jorge, Huesca, Huesca
  - Hospital Clínico de Santiago, Santiago de Compostela, La Coruña
  - Hospital Universitario de Fuenlabrada, Fuenlabrada, Madrid
  - Hospital Universitario de La Princesa, Madrid, Madrid
  - Hospital Universitario La Paz, Madrid, Madrid
  - Hospital Universitario de Torrejón, Torrejón de Ardoz, Madrid
  - Hospital Universitario de Navarra, Pamplona, Navarre
  - Hospital Universitario Central de Asturias, Oviedo, Principality of Asturias
  - Hospital Universitario Virgen del Rocío, Seville, Sevilla
  - Hospital Universitario y Politécnico La Fe, Valencia, Valencia
  - Hospital Rio Hortega, Valladolid, Valladolid
  - Hospital Clínico Universitario de Valladolid, Valladolid, Valladolid
  - Hospital de Galdakao, Galdakao, Vizcaya

REFERENCES:
- [Background] Loftus EV Jr. Clinical epidemiology of inflammatory bowel disease: Incidence, prevalence, and environmental influences. Gastroenterology. 2004 May;126(6):1504-17. doi: 10.1053/j.gastro.2004.01.063. PMID 15168363
- [Background] M'Koma AE. Inflammatory bowel disease: an expanding global health problem. Clin Med Insights Gastroenterol. 2013 Aug 14;6:33-47. doi: 10.4137/CGast.S12731. eCollection 2013. PMID 24833941
- [Background] Ng SC, Shi HY, Hamidi N, Underwood FE, Tang W, Benchimol EI, Panaccione R, Ghosh S, Wu JCY, Chan FKL, Sung JJY, Kaplan GG. Worldwide incidence and prevalence of inflammatory bowel disease in the 21st century: a systematic review of population-based studies. Lancet. 2017 Dec 23;390(10114):2769-2778. doi: 10.1016/S0140-6736(17)32448-0. Epub 2017 Oct 16. PMID 29050646
- [Background] Niewiadomski O, Studd C, Hair C, Wilson J, McNeill J, Knight R, Prewett E, Dabkowski P, Dowling D, Alexander S, Allen B, Tacey M, Connell W, Desmond P, Bell S. Health Care Cost Analysis in a Population-based Inception Cohort of Inflammatory Bowel Disease Patients in the First Year of Diagnosis. J Crohns Colitis. 2015 Nov;9(11):988-96. doi: 10.1093/ecco-jcc/jjv117. Epub 2015 Jun 30. PMID 26129692
- [Background] Bewtra M, Su C, Lewis JD. Trends in hospitalization rates for inflammatory bowel disease in the United States. Clin Gastroenterol Hepatol. 2007 May;5(5):597-601. doi: 10.1016/j.cgh.2007.01.015. Epub 2007 Mar 26. PMID 17382602
- [Background] Colombel JF, Sandborn WJ, Reinisch W, Mantzaris GJ, Kornbluth A, Rachmilewitz D, Lichtiger S, D'Haens G, Diamond RH, Broussard DL, Tang KL, van der Woude CJ, Rutgeerts P; SONIC Study Group. Infliximab, azathioprine, or combination therapy for Crohn's disease. N Engl J Med. 2010 Apr 15;362(15):1383-95. doi: 10.1056/NEJMoa0904492. PMID 20393175
- [Background] Gisbert JP, Marin AC, Chaparro M. The Risk of Relapse after Anti-TNF Discontinuation in Inflammatory Bowel Disease: Systematic Review and Meta-Analysis. Am J Gastroenterol. 2016 May;111(5):632-47. doi: 10.1038/ajg.2016.54. Epub 2016 Mar 22. PMID 27002797
- [Background] Gisbert JP, Domenech E. [Vedolizumab in the treatment of Crohn's disease]. Gastroenterol Hepatol. 2015 May;38(5):338-48. doi: 10.1016/j.gastrohep.2014.12.003. Epub 2015 Jan 23. Spanish. PMID 25619903
- [Background] Domenech E, Gisbert JP. Efficacy and safety of vedolizumab in the treatment of ulcerative colitis. Gastroenterol Hepatol. 2016 Dec;39(10):677-686. doi: 10.1016/j.gastrohep.2015.11.010. Epub 2016 Mar 2. English, Spanish. PMID 26948838
- [Background] Gisbert JP, Chaparro M. Ustekinumab to treat Crohn's disease. Gastroenterol Hepatol. 2017 Dec;40(10):688-698. doi: 10.1016/j.gastrohep.2017.08.006. Epub 2017 Oct 16. English, Spanish. PMID 29042094
- [Background] Ford AC, Sandborn WJ, Khan KJ, Hanauer SB, Talley NJ, Moayyedi P. Efficacy of biological therapies in inflammatory bowel disease: systematic review and meta-analysis. Am J Gastroenterol. 2011 Apr;106(4):644-59, quiz 660. doi: 10.1038/ajg.2011.73. Epub 2011 Mar 15. PMID 21407183
- [Background] Stidham RW, Lee TC, Higgins PD, Deshpande AR, Sussman DA, Singal AG, Elmunzer BJ, Saini SD, Vijan S, Waljee AK. Systematic review with network meta-analysis: the efficacy of anti-TNF agents for the treatment of Crohn's disease. Aliment Pharmacol Ther. 2014 Jun;39(12):1349-62. doi: 10.1111/apt.12749. Epub 2014 Apr 20. PMID 24749763
- [Background] Gordon JP, McEwan PC, Maguire A, Sugrue DM, Puelles J. Characterizing unmet medical need and the potential role of new biologic treatment options in patients with ulcerative colitis and Crohn's disease: a systematic review and clinician surveys. Eur J Gastroenterol Hepatol. 2015 Jul;27(7):804-12. doi: 10.1097/MEG.0000000000000378. PMID 25933126
- [Background] Ding NS, Hart A, De Cruz P. Systematic review: predicting and optimising response to anti-TNF therapy in Crohn's disease - algorithm for practical management. Aliment Pharmacol Ther. 2016 Jan;43(1):30-51. doi: 10.1111/apt.13445. Epub 2015 Oct 30. PMID 26515897
- [Background] Park SH, Aniwan S, Loftus EV Jr. Advances in the use of biologics and other novel drugs for managing inflammatory bowel disease. Curr Opin Pharmacol. 2017 Dec;37:65-71. doi: 10.1016/j.coph.2017.09.007. Epub 2017 Oct 6. PMID 28992449
- [Background] Lopetuso LR, Gerardi V, Papa V, Scaldaferri F, Rapaccini GL, Gasbarrini A, Papa A. Can We Predict the Efficacy of Anti-TNF-alpha Agents? Int J Mol Sci. 2017 Sep 14;18(9):1973. doi: 10.3390/ijms18091973. PMID 28906475
- [Background] Siegel CA, Melmed GY. Predicting response to Anti-TNF Agents for the treatment of crohn's disease. Therap Adv Gastroenterol. 2009 Jul;2(4):245-51. doi: 10.1177/1756283X09336364. PMID 21180547
- [Background] Kopylov U, Seidman E. Predicting durable response or resistance to antitumor necrosis factor therapy in inflammatory bowel disease. Therap Adv Gastroenterol. 2016 Jul;9(4):513-26. doi: 10.1177/1756283X16638833. Epub 2016 Apr 1. PMID 27366220
- [Background] Hindryckx P, Vande Casteele N, Novak G, Khanna R, D'Haens G, Sandborn WJ, Danese S, Jairath V, Feagan BG. The Expanding Therapeutic Armamentarium for Inflammatory Bowel Disease: How to Choose the Right Drug[s] for Our Patients? J Crohns Colitis. 2018 Jan 5;12(1):105-119. doi: 10.1093/ecco-jcc/jjx117. PMID 28961959
- [Background] Tew GW, Hackney JA, Gibbons D, Lamb CA, Luca D, Egen JG, Diehl L, Eastham Anderson J, Vermeire S, Mansfield JC, Feagan BG, Panes J, Baumgart DC, Schreiber S, Dotan I, Sandborn WJ, Kirby JA, Irving PM, De Hertogh G, Van Assche GA, Rutgeerts P, O'Byrne S, Hayday A, Keir ME. Association Between Response to Etrolizumab and Expression of Integrin alphaE and Granzyme A in Colon Biopsies of Patients With Ulcerative Colitis. Gastroenterology. 2016 Feb;150(2):477-87.e9. doi: 10.1053/j.gastro.2015.10.041. Epub 2015 Oct 30. PMID 26522261
- [Background] Dahlen R, Magnusson MK, Bajor A, Lasson A, Ung KA, Strid H, Ohman L. Global mucosal and serum cytokine profile in patients with ulcerative colitis undergoing anti-TNF therapy. Scand J Gastroenterol. 2015;50(9):1118-26. doi: 10.3109/00365521.2015.1031167. Epub 2015 Apr 16. PMID 25877762
- [Background] Eftekhari P, Glaubitz L, Breidert M, Neurath MF, Atreya R. Physiological intermolecular modification spectroscopy for the prediction of response to anti-tumor necrosis factor therapy in patients with inflammatory bowel diseases. Dig Dis. 2014;32(4):446-54. doi: 10.1159/000358151. Epub 2014 Jun 23. PMID 24969293
- [Background] Meuwis MA, Fillet M, Lutteri L, Maree R, Geurts P, de Seny D, Malaise M, Chapelle JP, Wehenkel L, Belaiche J, Merville MP, Louis E. Proteomics for prediction and characterization of response to infliximab in Crohn's disease: a pilot study. Clin Biochem. 2008 Aug;41(12):960-7. doi: 10.1016/j.clinbiochem.2008.04.021. Epub 2008 May 6. PMID 18489908
- [Background] Hassan EA, Ramadan HK, Ismael AA, Mohamed KF, El-Attar MM, Alhelali I. Noninvasive biomarkers as surrogate predictors of clinical and endoscopic remission after infliximab induction in patients with refractory ulcerative colitis. Saudi J Gastroenterol. 2017 Jul-Aug;23(4):238-245. doi: 10.4103/sjg.SJG_599_16. PMID 28721978
- [Background] Feng T, Chen B, Li L, Huang S, Ben-Horin S, Qiu Y, Feng R, Li M, Mao R, He Y, Zeng Z, Zhang S, Chen M. Serum Interleukin 9 Levels Predict Disease Severity and the Clinical Efficacy of Infliximab in Patients with Crohn's Disease. Inflamm Bowel Dis. 2017 Oct;23(10):1817-1824. doi: 10.1097/MIB.0000000000001172. PMID 28644181
- [Background] Fuchs F, Schillinger D, Atreya R, Hirschmann S, Fischer S, Neufert C, Atreya I, Neurath MF, Zundler S. Clinical Response to Vedolizumab in Ulcerative Colitis Patients Is Associated with Changes in Integrin Expression Profiles. Front Immunol. 2017 Jul 3;8:764. doi: 10.3389/fimmu.2017.00764. eCollection 2017. PMID 28717358
- [Background] Planell N, Masamunt MC, Leal RF, Rodriguez L, Esteller M, Lozano JJ, Ramirez A, Ayrizono MLS, Coy CSR, Alfaro I, Ordas I, Visvanathan S, Ricart E, Guardiola J, Panes J, Salas A. Usefulness of Transcriptional Blood Biomarkers as a Non-invasive Surrogate Marker of Mucosal Healing and Endoscopic Response in Ulcerative Colitis. J Crohns Colitis. 2017 Oct 27;11(11):1335-1346. doi: 10.1093/ecco-jcc/jjx091. PMID 28981629
- [Background] Barcelo-Batllori S, Andre M, Servis C, Levy N, Takikawa O, Michetti P, Reymond M, Felley-Bosco E. Proteomic analysis of cytokine induced proteins in human intestinal epithelial cells: implications for inflammatory bowel diseases. Proteomics. 2002 May;2(5):551-60. doi: 10.1002/1615-9861(200205)2:53.0.CO;2-O. PMID 11987129
- [Background] Han NY, Choi W, Park JM, Kim EH, Lee H, Hahm KB. Label-free quantification for discovering novel biomarkers in the diagnosis and assessment of disease activity in inflammatory bowel disease. J Dig Dis. 2013 Apr;14(4):166-74. doi: 10.1111/1751-2980.12035. PMID 23320753
- [Background] Hardwidge PR, Rodriguez-Escudero I, Goode D, Donohoe S, Eng J, Goodlett DR, Aebersold R, Finlay BB. Proteomic analysis of the intestinal epithelial cell response to enteropathogenic Escherichia coli. J Biol Chem. 2004 May 7;279(19):20127-36. doi: 10.1074/jbc.M401228200. Epub 2004 Feb 26. PMID 14988394
- [Background] Hsieh SY, Shih TC, Yeh CY, Lin CJ, Chou YY, Lee YS. Comparative proteomic studies on the pathogenesis of human ulcerative colitis. Proteomics. 2006 Oct;6(19):5322-31. doi: 10.1002/pmic.200500541. PMID 16947118
- [Background] M'Koma AE, Seeley EH, Washington MK, Schwartz DA, Muldoon RL, Herline AJ, Wise PE, Caprioli RM. Proteomic profiling of mucosal and submucosal colonic tissues yields protein signatures that differentiate the inflammatory colitides. Inflamm Bowel Dis. 2011 Apr;17(4):875-83. doi: 10.1002/ibd.21442. Epub 2010 Aug 30. PMID 20806340
- [Background] Nanni P, Mezzanotte L, Roda G, Caponi A, Levander F, James P, Roda A. Differential proteomic analysis of HT29 Cl.16E and intestinal epithelial cells by LC ESI/QTOF mass spectrometry. J Proteomics. 2009 Jul 21;72(5):865-73. doi: 10.1016/j.jprot.2008.12.010. Epub 2009 Jan 8. PMID 19168159
- [Background] Presley LL, Ye J, Li X, Leblanc J, Zhang Z, Ruegger PM, Allard J, McGovern D, Ippoliti A, Roth B, Cui X, Jeske DR, Elashoff D, Goodglick L, Braun J, Borneman J. Host-microbe relationships in inflammatory bowel disease detected by bacterial and metaproteomic analysis of the mucosal-luminal interface. Inflamm Bowel Dis. 2012 Mar;18(3):409-17. doi: 10.1002/ibd.21793. Epub 2011 Jun 22. PMID 21698720
- [Background] Seeley EH, Washington MK, Caprioli RM, M'Koma AE. Proteomic patterns of colonic mucosal tissues delineate Crohn's colitis and ulcerative colitis. Proteomics Clin Appl. 2013 Aug;7(7-8):541-9. doi: 10.1002/prca.201200107. Epub 2013 May 8. PMID 23382084
- [Background] Shkoda A, Werner T, Daniel H, Gunckel M, Rogler G, Haller D. Differential protein expression profile in the intestinal epithelium from patients with inflammatory bowel disease. J Proteome Res. 2007 Mar;6(3):1114-25. doi: 10.1021/pr060433m. PMID 17330946
- [Background] Nanni P, Parisi D, Roda G, Casale M, Belluzzi A, Roda E, Mayer L, Roda A. Serum protein profiling in patients with inflammatory bowel diseases using selective solid-phase bulk extraction, matrix-assisted laser desorption/ionization time-of-flight mass spectrometry and chemometric data analysis. Rapid Commun Mass Spectrom. 2007;21(24):4142-8. doi: 10.1002/rcm.3323. PMID 18022963
- [Background] Arbelaiz A, Azkargorta M, Krawczyk M, Santos-Laso A, Lapitz A, Perugorria MJ, Erice O, Gonzalez E, Jimenez-Aguero R, Lacasta A, Ibarra C, Sanchez-Campos A, Jimeno JP, Lammert F, Milkiewicz P, Marzioni M, Macias RIR, Marin JJG, Patel T, Gores GJ, Martinez I, Elortza F, Falcon-Perez JM, Bujanda L, Banales JM. Serum extracellular vesicles contain protein biomarkers for primary sclerosing cholangitis and cholangiocarcinoma. Hepatology. 2017 Oct;66(4):1125-1143. doi: 10.1002/hep.29291. Epub 2017 Aug 26. PMID 28555885
- [Background] Spitzer MH, Nolan GP. Mass Cytometry: Single Cells, Many Features. Cell. 2016 May 5;165(4):780-91. doi: 10.1016/j.cell.2016.04.019. PMID 27153492
- [Background] Bendall SC, Nolan GP, Roederer M, Chattopadhyay PK. A deep profiler's guide to cytometry. Trends Immunol. 2012 Jul;33(7):323-32. doi: 10.1016/j.it.2012.02.010. Epub 2012 Apr 2. PMID 22476049
- [Background] Stikvoort A, Chen Y, Radestad E, Torlen J, Lakshmikanth T, Bjorklund A, Mikes J, Achour A, Gertow J, Sundberg B, Remberger M, Sundin M, Mattsson J, Brodin P, Uhlin M. Combining Flow and Mass Cytometry in the Search for Biomarkers in Chronic Graft-versus-Host Disease. Front Immunol. 2017 Jun 19;8:717. doi: 10.3389/fimmu.2017.00717. eCollection 2017. PMID 28674539
- [Background] Nair N, Mei HE, Chen SY, Hale M, Nolan GP, Maecker HT, Genovese M, Fathman CG, Whiting CC. Mass cytometry as a platform for the discovery of cellular biomarkers to guide effective rheumatic disease therapy. Arthritis Res Ther. 2015 May 18;17(1):127. doi: 10.1186/s13075-015-0644-z. PMID 25981462
- [Background] Gaudilliere B, Fragiadakis GK, Bruggner RV, Nicolau M, Finck R, Tingle M, Silva J, Ganio EA, Yeh CG, Maloney WJ, Huddleston JI, Goodman SB, Davis MM, Bendall SC, Fantl WJ, Angst MS, Nolan GP. Clinical recovery from surgery correlates with single-cell immune signatures. Sci Transl Med. 2014 Sep 24;6(255):255ra131. doi: 10.1126/scitranslmed.3009701. PMID 25253674
- [Background] Fergusson JR, Smith KE, Fleming VM, Rajoriya N, Newell EW, Simmons R, Marchi E, Bjorkander S, Kang YH, Swadling L, Kurioka A, Sahgal N, Lockstone H, Baban D, Freeman GJ, Sverremark-Ekstrom E, Davis MM, Davenport MP, Venturi V, Ussher JE, Willberg CB, Klenerman P. CD161 defines a transcriptional and functional phenotype across distinct human T cell lineages. Cell Rep. 2014 Nov 6;9(3):1075-88. doi: 10.1016/j.celrep.2014.09.045. Epub 2014 Oct 23. PMID 25437561
- [Background] van Unen V, Li N, Molendijk I, Temurhan M, Hollt T, van der Meulen-de Jong AE, Verspaget HW, Mearin ML, Mulder CJ, van Bergen J, Lelieveldt BP, Koning F. Mass Cytometry of the Human Mucosal Immune System Identifies Tissue- and Disease-Associated Immune Subsets. Immunity. 2016 May 17;44(5):1227-39. doi: 10.1016/j.immuni.2016.04.014. Epub 2016 May 10. PMID 27178470
- [Background] Gerich ME, McGovern DP. Towards personalized care in IBD. Nat Rev Gastroenterol Hepatol. 2014 May;11(5):287-99. doi: 10.1038/nrgastro.2013.242. Epub 2013 Dec 17. PMID 24345887
- [Background] Peyrin-Biroulet L, Sandborn W, Sands BE, Reinisch W, Bemelman W, Bryant RV, D'Haens G, Dotan I, Dubinsky M, Feagan B, Fiorino G, Gearry R, Krishnareddy S, Lakatos PL, Loftus EV Jr, Marteau P, Munkholm P, Murdoch TB, Ordas I, Panaccione R, Riddell RH, Ruel J, Rubin DT, Samaan M, Siegel CA, Silverberg MS, Stoker J, Schreiber S, Travis S, Van Assche G, Danese S, Panes J, Bouguen G, O'Donnell S, Pariente B, Winer S, Hanauer S, Colombel JF. Selecting Therapeutic Targets in Inflammatory Bowel Disease (STRIDE): Determining Therapeutic Goals for Treat-to-Target. Am J Gastroenterol. 2015 Sep;110(9):1324-38. doi: 10.1038/ajg.2015.233. Epub 2015 Aug 25. PMID 26303131
- [Background] Rieder F, Karrasch T, Ben-Horin S, Schirbel A, Ehehalt R, Wehkamp J, de Haar C, Velin D, Latella G, Scaldaferri F, Rogler G, Higgins P, Sans M. Results of the 2nd scientific workshop of the ECCO (III): basic mechanisms of intestinal healing. J Crohns Colitis. 2012 Apr;6(3):373-85. doi: 10.1016/j.crohns.2011.11.009. Epub 2011 Dec 11. PMID 22405177
- [Background] Neurath MF, Travis SP. Mucosal healing in inflammatory bowel diseases: a systematic review. Gut. 2012 Nov;61(11):1619-35. doi: 10.1136/gutjnl-2012-302830. Epub 2012 Jul 27. PMID 22842618
- [Background] Khanna R, Bouguen G, Feagan BG, D'Haens G, Sandborn WJ, Dubcenco E, Baker KA, Levesque BG. A systematic review of measurement of endoscopic disease activity and mucosal healing in Crohn's disease: recommendations for clinical trial design. Inflamm Bowel Dis. 2014 Oct;20(10):1850-61. doi: 10.1097/MIB.0000000000000131. PMID 25029615
- [Background] Colombel JF, Rutgeerts P, Reinisch W, Esser D, Wang Y, Lang Y, Marano CW, Strauss R, Oddens BJ, Feagan BG, Hanauer SB, Lichtenstein GR, Present D, Sands BE, Sandborn WJ. Early mucosal healing with infliximab is associated with improved long-term clinical outcomes in ulcerative colitis. Gastroenterology. 2011 Oct;141(4):1194-201. doi: 10.1053/j.gastro.2011.06.054. Epub 2011 Jun 30. PMID 21723220
- [Background] Peyrin-Biroulet L, Ferrante M, Magro F, Campbell S, Franchimont D, Fidder H, Strid H, Ardizzone S, Veereman-Wauters G, Chevaux JB, Allez M, Danese S, Sturm A; Scientific Committee of the European Crohn's and Colitis Organization. Results from the 2nd Scientific Workshop of the ECCO. I: Impact of mucosal healing on the course of inflammatory bowel disease. J Crohns Colitis. 2011 Oct;5(5):477-83. doi: 10.1016/j.crohns.2011.06.009. Epub 2011 Aug 3. PMID 21939925
- [Background] Shah SC, Colombel JF, Sands BE, Narula N. Systematic review with meta-analysis: mucosal healing is associated with improved long-term outcomes in Crohn's disease. Aliment Pharmacol Ther. 2016 Feb;43(3):317-33. doi: 10.1111/apt.13475. Epub 2015 Nov 25. PMID 26607562
- [Background] Pineton de Chambrun G, Blanc P, Peyrin-Biroulet L. Current evidence supporting mucosal healing and deep remission as important treatment goals for inflammatory bowel disease. Expert Rev Gastroenterol Hepatol. 2016 Aug;10(8):915-27. doi: 10.1586/17474124.2016.1174064. Epub 2016 Apr 18. PMID 27043489
- [Background] Scoville EA, Schwartz DA. Endoscopy in inflammatory bowel disease: advances in disease management. Gastrointest Endosc. 2017 Dec;86(6):952-961. doi: 10.1016/j.gie.2017.08.034. Epub 2017 Sep 6. No abstract available. PMID 28886962
- [Background] Arijs I, Li K, Toedter G, Quintens R, Van Lommel L, Van Steen K, Leemans P, De Hertogh G, Lemaire K, Ferrante M, Schnitzler F, Thorrez L, Ma K, Song XY, Marano C, Van Assche G, Vermeire S, Geboes K, Schuit F, Baribaud F, Rutgeerts P. Mucosal gene signatures to predict response to infliximab in patients with ulcerative colitis. Gut. 2009 Dec;58(12):1612-9. doi: 10.1136/gut.2009.178665. Epub 2009 Aug 20. PMID 19700435
- [Background] Arijs I, Quintens R, Van Lommel L, Van Steen K, De Hertogh G, Lemaire K, Schraenen A, Perrier C, Van Assche G, Vermeire S, Geboes K, Schuit F, Rutgeerts P. Predictive value of epithelial gene expression profiles for response to infliximab in Crohn's disease. Inflamm Bowel Dis. 2010 Dec;16(12):2090-8. doi: 10.1002/ibd.21301. PMID 20848504
- [Background] Li Z, Arijs I, De Hertogh G, Vermeire S, Noman M, Bullens D, Coorevits L, Sagaert X, Schuit F, Rutgeerts P, Ceuppens JL, Van Assche G. Reciprocal changes of Foxp3 expression in blood and intestinal mucosa in IBD patients responding to infliximab. Inflamm Bowel Dis. 2010 Aug;16(8):1299-310. doi: 10.1002/ibd.21229. PMID 20196149
- [Background] Olsen T, Goll R, Cui G, Christiansen I, Florholmen J. TNF-alpha gene expression in colorectal mucosa as a predictor of remission after induction therapy with infliximab in ulcerative colitis. Cytokine. 2009 May;46(2):222-7. doi: 10.1016/j.cyto.2009.02.001. Epub 2009 Mar 14. PMID 19286392
- [Background] Rismo R, Olsen T, Cui G, Christiansen I, Florholmen J, Goll R. Mucosal cytokine gene expression profiles as biomarkers of response to infliximab in ulcerative colitis. Scand J Gastroenterol. 2012 May;47(5):538-47. doi: 10.3109/00365521.2012.667146. PMID 22486187
- [Background] Viazis N, Giakoumis M, Bamias G, Goukos D, Koukouratos T, Katopodi K, Karatzas P, Triantos C, Tsolias C, Theocharis G, Daikos GL, Ladas SD, Karamanolis DG, Mantzaris GJ. Predictors of tissue healing in ulcerative colitis patients treated with anti-TNF. Dig Liver Dis. 2017 Jan;49(1):29-33. doi: 10.1016/j.dld.2016.10.008. Epub 2016 Oct 20. PMID 27866814
- [Background] D'Haens G, Sandborn WJ, Feagan BG, Geboes K, Hanauer SB, Irvine EJ, Lemann M, Marteau P, Rutgeerts P, Scholmerich J, Sutherland LR. A review of activity indices and efficacy end points for clinical trials of medical therapy in adults with ulcerative colitis. Gastroenterology. 2007 Feb;132(2):763-86. doi: 10.1053/j.gastro.2006.12.038. Epub 2006 Dec 20. No abstract available. PMID 17258735
- [Background] Daperno M, D'Haens G, Van Assche G, Baert F, Bulois P, Maunoury V, Sostegni R, Rocca R, Pera A, Gevers A, Mary JY, Colombel JF, Rutgeerts P. Development and validation of a new, simplified endoscopic activity score for Crohn's disease: the SES-CD. Gastrointest Endosc. 2004 Oct;60(4):505-12. doi: 10.1016/s0016-5107(04)01878-4. PMID 15472670
- [Background] Vuitton L, Marteau P, Sandborn WJ, Levesque BG, Feagan B, Vermeire S, Danese S, D'Haens G, Lowenberg M, Khanna R, Fiorino G, Travis S, Mary JY, Peyrin-Biroulet L. IOIBD technical review on endoscopic indices for Crohn's disease clinical trials. Gut. 2016 Sep;65(9):1447-55. doi: 10.1136/gutjnl-2015-309903. Epub 2015 Sep 9. PMID 26353983
- [Background] Kamm MA, Sandborn WJ, Gassull M, Schreiber S, Jackowski L, Butler T, Lyne A, Stephenson D, Palmen M, Joseph RE. Once-daily, high-concentration MMX mesalamine in active ulcerative colitis. Gastroenterology. 2007 Jan;132(1):66-75; quiz 432-3. doi: 10.1053/j.gastro.2006.10.011. Epub 2006 Oct 12. PMID 17241860
- [Background] D'Haens GR, Panaccione R, Higgins PD, Vermeire S, Gassull M, Chowers Y, Hanauer SB, Herfarth H, Hommes DW, Kamm M, Lofberg R, Quary A, Sands B, Sood A, Watermeyer G, Lashner B, Lemann M, Plevy S, Reinisch W, Schreiber S, Siegel C, Targan S, Watanabe M, Feagan B, Sandborn WJ, Colombel JF, Travis S. The London Position Statement of the World Congress of Gastroenterology on Biological Therapy for IBD with the European Crohn's and Colitis Organization: when to start, when to stop, which drug to choose, and how to predict response? Am J Gastroenterol. 2011 Feb;106(2):199-212; quiz 213. doi: 10.1038/ajg.2010.392. Epub 2010 Nov 2. PMID 21045814
- [Background] Van Assche G, Sandborn WJ, Feagan BG, Salzberg BA, Silvers D, Monroe PS, Pandak WM, Anderson FH, Valentine JF, Wild GE, Geenen DJ, Sprague R, Targan SR, Rutgeerts P, Vexler V, Young D, Shames RS. Daclizumab, a humanised monoclonal antibody to the interleukin 2 receptor (CD25), for the treatment of moderately to severely active ulcerative colitis: a randomised, double blind, placebo controlled, dose ranging trial. Gut. 2006 Nov;55(11):1568-74. doi: 10.1136/gut.2005.089854. Epub 2006 Apr 7. PMID 16603634
- [Background] D'Haens G, Feagan B, Colombel JF, Sandborn WJ, Reinisch W, Rutgeerts P, Carbonnel F, Mary JY, Danese S, Fedorak RN, Hanauer S, Lemann M; International Organization for Inflammatory Bowel Diseases (IOIBD) and the Clinical Trial Committee Clincom of the European Crohn's and Colitis Organisation (ECCO). Challenges to the design, execution, and analysis of randomized controlled trials for inflammatory bowel disease. Gastroenterology. 2012 Dec;143(6):1461-9. doi: 10.1053/j.gastro.2012.09.031. Epub 2012 Sep 20. PMID 23000597
- [Background] Nunes T, Barreiro-de Acosta M, Nos P, Marin-Jimenez I, Bermejo F, Ceballos D, Iglesias E, Gomez-Senent S, Torres Y, Ponferrada A, Arevalo JA, Hernandez V, Calvet X, Ginard D, Monfort D, Chaparro M, Mancenido N, Dominguez-Antonaya M, Villalon C, Perez-Calle JL, Munoz C, Nunez H, Carpio D, Aramendiz R, Bujanda L, Estrada-Oncins S, Hermida C, Barrio J, Casis MB, Duenas-Sadornil MC, Fernandez L, Calvo-Cenizo MM, Botella B, de Francisco R, Ayala E, Sans M; RECLICU Study Group of GETECCU. Usefulness of oral beclometasone dipropionate in the treatment of active ulcerative colitis in clinical practice: the RECLICU Study. J Crohns Colitis. 2010 Dec;4(6):629-36. doi: 10.1016/j.crohns.2010.07.003. PMID 21122572